CLINICAL TRIAL: NCT04561323
Title: Dual-energy CT in the Diagnosis of All-Cause Acute Bowel Ischemia
Brief Title: Diagnosing Acute Onset Insufficient Intestinal Blood Flow (Bowel Ischemia) With a Novel CT Technique Called Dual-energy CT (DECT). This Observational Study Seeks to Evaluate Whether DECT Can Improve the Diagnosis of Bowel Ischemia and How the DECT Findings Correlate With Intraoperative Findings
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jack Xu, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-20029655
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Bowel Ischemia; Acute Bowel Ischemia / Infarction
Keywords: Dual-energy CT
MeSH Terms: conditions — Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dual-energy CT — Patients suspected of acute bowel ischemia will be scanned in the dual-energy CT scanner.
  The abdominal imaging protocols are predetermined by the Department of Diagnostic Radiology, Righospitalet, Denmark.

SUMMARY:
The aim of this study is to evaluate the performance of dual-energy CT (DECT) in the diagnosis of acute bowel ischemia (ABI). ABI is a condition characterised by inadequate blood supply to portions of the intestine. ABI is a relatively rare condition, but is associated with a high mortality rate.

DECT is an emerging field within radiology. Few reports have reported an increased conspicuity for ABI using DECT compared with conventional CT, which is the current preoperative golden standard.

The investigators hypothesize that DECT increases conspicuity of ABI compared with conventional CT and that DECT image findings correlate with the intraoperative findings.

ELIGIBILITY:
Inclusion Criteria:

* Referred on the suspicion of acute bowel ischemia

Exclusion Criteria:

* Patient not scanned with DECT
* Patient does not undergo abdominal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists of admitted patients at Rigshospitalet, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Adding DECT information increases assessor confidence without lowering the specificity compared with standard CT in the diagnosis and/or exclusion of ABI. | 10 minutes

SECONDARY OUTCOMES:
Intraoperative ICG fluorescence angiogram perfusion assessment and its correlation to DECT image evaluation. | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Diagnostic Radiology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No